CLINICAL TRIAL: NCT06325930
Title: An Open-Label Phase 1 Study in Healthy Adult Male Subjects to Investigate the Absorption, Metabolism, and Excretion of [14C]-HU6 Following Single-Dose Oral Administration
Brief Title: A Study to Investigate the Absorption, Metabolism, and Excretion of [14C]-HU6
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rivus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RIV-HU6-105
Record Dates: First submitted 2024-03-13; First posted 2024-03-22 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-04

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- single dose of [14C]-HU6 (Experimental)
  Interventions: Drug: [14C]-HU6

INTERVENTIONS:
Drug: [14C]-HU6 — [14C]-HU6 following a single dose of HU6 in healthy, adult male subjects

SUMMARY:
This is a single-center, non-randomized, open-label Phase 1 study to characterize the absorption, metabolism, excretion, mass balance, pharmacokinetics (PK), safety and tolerability of HU6 following administration of a single dose of [14C]-HU6 in a fed state with a standard meal administered approximately 15 minutes prior to dosing.

DETAILED DESCRIPTION:
This is a single-center, non-randomized, open-label Phase 1 study to characterize the absorption, metabolism, excretion, mass balance, pharmacokinetics (PK), safety and tolerability of HU6 following administration of a single dose of [14C]-HU6 in a fed state with a standard meal administered approximately 15 minutes prior to dosing.

Healthy, adult males aged 18 to 55, inclusive, who have provided written informed consent, will be screened, and subjects who meet all eligibility criteria may be enrolled into the study within 28 days of Screening.

Approximately 8 eligible subjects will be admitted on Day -1, and baseline assessments will be completed. On Day 1, 8 subjects will receive a single dose of [14C]-HU6 in a fed state. If ≥ 85% (mean of all subjects) of the 14C label has been recovered in samples collected and analyzed through 336 hours after dosing and the mean of individual 14C recovery is < 1% on each of 2 consecutive days, all subjects will be discharged from the Pharmaron Clinical Pharmacology Center (CPC) on Day 15 after completion of all 336-hour timepoint assessments.

ELIGIBILITY:
Inclusion Criteria:

* Capable of understanding the written informed consent form (ICF), willingly provide valid, signed written informed consent and willing and able to comply with the schedule, requirements and restrictions of the study
* Healthy males between 18.0 and 55.0 years of age (inclusive) at the time of Screening.
* Body mass index (BMI) ≥ 18.0 kg/m2 and ≤ 32.5 kg/m2 at Screening; body weight ≥ 55.0 kg and ≤ 100.0 kg at Screening.
* Considered to be in good health by the Investigator, as determined by medical history, physical examination, vital signs (VS) measurements, 12-lead electrocardiogram (ECG), and clinical laboratory test results.
* Male subjects with female sexual partner(s) of reproductive potential may be enrolled if the male:

  1. is documented to be surgically sterile (i.e., successfully vasectomized), or
  2. agrees to use 2 methods of highly effective contraception (e.g, condom plus spermicide) and female partner's use of a reliable form of contraception during intercourse for the duration of the study, and for at least 90 days after receiving study drug and agrees to refrain from sperm donation from the time of Screening through 90 days post dose.

Exclusion Criteria:

* History or presence of any condition (e.g., chronic diarrhea), gastrointestinal bleeding, including related to hemorrhoids or prior surgery (e.g., gastric bypass) that, in the opinion of the Investigator, poses a significant risk to subject safety and/or achievement of study objectives.
* History of cancer that has not been in complete remission for > 5 years (except basal cell skin cancer or squamous cell skin cancer with a history of curative treatment and no recurrence for > 1 year prior to Screening), as judged by the Investigator.
* Acute illness within 14 days prior to study drug administration on Day 1, unless mild in severity and enrollment is approved by both the Investigator and Sponsor's medical representative.
* History of COVID symptoms or positive COVID test within 2 weeks prior to admission date.
* Any history of serious allergic drug reactions.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2024-03-26 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-05-07 (Actual)

PRIMARY OUTCOMES:
To assess the mass balance | Up to Day 29
  (i.e., the cumulative excretion of total 14C in urine and feces), of [14C]-HU6 following a single dose of [14C]-HU6, in healthy, adult male subjects

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmaron Clinical Pharmacology Center (CPC), Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No